CLINICAL TRIAL: NCT03879278
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of NPT189 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Mild infusion reactions were observed in two healthy volunteers.
Sponsor: Proclara Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPT189-CL002
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-03

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Immunoglobulin G

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment 2 mg/kg (Other): Five IV doses of 2 mg/kg NPT189 (n = 6) or matching placebo (n = 2) administered once per week
  Interventions: Drug: NPT189
- Treatment 5 mg/kg (Other): Five IV doses of 5 mg/kg NPT189 (n = 6) or matching placebo (n = 2) administered once per week
  Interventions: Drug: NPT189
- Treatment 12.5 mg/kg (Other): Five IV doses of 12.5 mg/kg NPT189 (n = 6) or matching placebo (n = 2) administered once per week
  Interventions: Drug: NPT189

INTERVENTIONS:
Drug: NPT189 — NPT189 is a recombinant immunoglobulin Fc fusion of GAIM (GAIM-IgG1Fc) as a potential treatment for peripheral amyloidosis.
  Other Names: IgG1 (Immunoglobulin G); Fusion Protein; GAIM (General Amyloid Interaction Motif)

SUMMARY:
This will be a Phase 1, randomized, double-blind, single center, placebo-controlled, multiple ascending dose (MAD) study in a maximum of 3 cohorts of 8 healthy male and female subjects each. Subjects in Cohorts 1, 2 and 3 will receive ascending multiple IV doses of NPT189 or matching placebo.

DETAILED DESCRIPTION:
This study is a Phase 1, randomized, double-blind, placebo-controlled, multiple dose, dose escalation safety, tolerability and PK study of NPT189 in healthy subjects. Three dose cohorts are planned each with a maximum of 8 subjects (6 active: 2 placebo) enrolled per cohort. Eligible subjects will be administered NPT189 by IV infusions at the dose specified for their cohort (i.e., 2 mg/kg, 5 mg/kg, and 12.5 mg/kg) or a matching placebo. Subjects will receive a total of 5 doses of NPT189, with doses administered at weekly intervals. Safety and tolerability will be assessed by analysis of adverse events (AEs), vital signs, electrocardiograms (ECG), laboratory and physical examinations. PK will be assessed by analysis of serum NPT189 concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years, inclusive, at screening
2. Weight 45-120 kg, inclusive
3. Body Mass Index of 18.0-32.0 kg/m2, inclusive
4. Female subjects of childbearing potential (defined as not surgically sterile or at least 2 years postmenopausal confirmed by a Screening Follicular Stimulating Hormone level of > 40) must agree to use two of the following forms of contraception from 60 days prior through 90 days following the dose of study drug: hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), IUD, complete abstinence, or vasectomized partner (6 months minimum) or male subjects who are sexually active with women of childbearing potential must agree to complete abstinence or to use a condom for 90 days following the dose of study drug.
5. No clinically significant abnormal findings on physical examination, vital signs, electrocardiogram (ECG), or clinical laboratory evaluation during screening; and systolic blood pressure between 140 mm and 90 mm Hg and diastolic blood pressure between 90 mm and 45 mm Hg.
6. Can understand and sign the informed consent document, can communicate with the Investigator, and can understand and comply with the requirements of the protocol.

Exclusion Criteria:

1. Have a past or present serious medical illness or other medical or social reason that in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Participation in a clinical trial (other than a screening visit) within 60 days of study drug administration.
3. Use of any over-the-counter or prescription medication , vitamin preparations and other food supplements, or herbal medications (e.g., St. John's Wort) within 14 days prior to the dose of study drug or during the study, with the exception of hormonal contraceptives for women of childbearing potential, unless approved by the Principal Investigator or use of beta-blockers within 30 days prior to dose of study drug or during the study.
4. Donation of blood or plasma within 30 days of the dose of study drug and throughout the duration of the study and for male subjects, donation of sperm through the duration of the study.
5. Women who are nursing, pregnant, suspected of being pregnant, or trying to become pregnant, or are lactating, have a positive serum pregnancy test at screening or urine pregnancy test prior to administration of study drug regardless of childbearing potential.
6. Positive blood screen for HIV, hepatitis B surface antigen (HbSAg), or hepatitis C as Screening, or a positive urine screen for alcohol (the day before each dose administration only) or, drugs of abuse, or cotinine at Screening and on the day before each dose administration.
7. Have clinically significant abnormalities in laboratory values as judged by the clinical investigator.
8. Have a history of alcoholism and/or drug abuse.
9. Unsuitable veins for infusion or blood sampling.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Adverse event assessment in subjects receiving multiple intravenous infusions of NPT189 | Day 1 through Day 112
  Summary of the frequency and percentage of adverse events

SECONDARY OUTCOMES:
Profile of pharmacokinetics (PK) of multiple intravenous (IV) infusions of NPT189 (Cmax) | Day 1 through Day 112
  Observed maximum concentration (Cmax)
Profile of pharmacokinetics (PK) of multiple intravenous (IV) infusions of NPT189 (Tmax) | Day 1 through Day 112
  Time of the maximum measured concentration (Tmax)
Profile of pharmacokinetics (PK) of multiple (IV) infusions of NPT189 (AUC 0-tau) | Day 1 through Day 112
  Area under the serum concentration-time curve over a dosing interval, tau
Profile of pharmacokinetics (PK) of multiple intravenous (IV) infusions of NPT189. Terminal elimination half-life (t 1/2) | Day 1 through DAy 112
  Terminal elimination half-life (t 1/2)
Profile of pharmacokinetics (PK) of multiple (IV) infusions of NPT189. Clearance (CL) | Day 1 through Day 112
  Clearance (CL)
Profile of pharmacokinetics (PK) of multiple (IV) infusions of NPT189. Volume of distribution (Vd) | Day 1 through Day 112
  Apparent volume of distribution (Vd)

CONTACTS AND LOCATIONS:
Overall Officials: Proclara Biosciences, Inc, Study Director — Proclara Biosciences
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No